CLINICAL TRIAL: NCT06672497
Title: Near Infrared Spectroscopy (NIRS) as a Method for Measuring Oxidative Capacity of Skeletal Muscle Mitochondria in Breast Cancer and All Gynecological Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: Furman University (Unknown); Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Jennifer Trilk, Professor of Biomedical Sciences and Director of the Human Performance Lab, University of South Carolina
Other Study IDs: 1853511
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Gynecologic Cancers; Mitochondrial Function
Keywords: nirs; mitochondrial oxidative capacity; muscle oxidative capacity; breast cancer; gynecological cancer; near infrared spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with breast or gynecological cancer and undergoing neoadjuvant chemotherapy.: Females ages 20...

SUMMARY:
Participants recruited for this study will be breast cancer or gynecological cancer patients who agree to participate in an exercise study examining the effects of chemotherapy on muscle mitochondrial oxidative capacity, a measure of skeletal muscle health. Participants will ride a stationary bicycle and the quadriceps muscle will be non-invasively evaluated.

DETAILED DESCRIPTION:
The NIRS participant testing will be performed in the University of South Carolina School of Medicine Greenville's Human Performance Laboratory located within Cancer Institute Faris Road facility. Testing will take approximately 30 minutes per session, with a maximum of 180 minutes of participation per patient. The independent variables in this study are drug regimen and number of chemotherapy treatments. The dependent variables in this study will be the change in oxygenation and deoxygenation status of the vastus lateralis as measured by the NIRS device, indicative of mitochondrial oxidative capacity, after a bout of cycling. Patients will be asked to avoid exercise and use of certain substances (tobacco, alcohol, caffeine, and contraindicated medications) 24 hours prior to testing.

Participants will be asked to perform exercise in shorts or equivalent. Participants will first sit at rest in a chair, as the NIRS device is applied to the vastus lateralis. The device will have double sided adhesive tape to lightly secure its position to the skin. The device will be wrapped in a black cloth to fully secure its position, limit device mobility, and block ambient light in the laboratory. Participants will then stand and walk to the cycle with the NIRS secured to the participant's leg. Participants will sit on the bike for a 2-minute rest while wearing a fitted mask that comfortably measures the participant's rate and amount of oxygen uptake (VO2) and other ventilatory measurements at rest and during exercise.

Researchers will determine the participant's lactate threshold curve and ventilatory threshold during a graded exercise test. The lactate threshold is a measure of the rate at which capillary blood lactate measurements rise as an effect of increased exercise intensity. The blood lactate curve will be used to determine an individualized power wattage for subsequent exercise testing of "on-off kinetics" (see below description). Capillary blood lactate levels will be obtained by finger stick for point of care testing. Ventilatory threshold will be measured using indirect calorimetry via a metabolic cart that captures expired gasses (O2 and CO2) through a comfortable silicone mask worn by the participant.

A baseline blood lactate level will be obtained at rest, then the participant will be instructed to cycle for three minutes beginning at 10W. After the 3-minute stage is complete, the power output will increase by 15 watts. The participant will cycle for 3 minutes at each stage until their lactate threshold reaches 4.0 mmol/L. Once the blood lactate reaches 4.0 mmol/L, one final, three-minute stage will be performed. A final lactate reading will be obtained at the completion of this exercise stage. The power output that is equivalent to 1.1x the wattage at which their lactate threshold exceeded 4.0 mmol/L will be used as the exercise intensity ("on-kinetics") for subsequent visits accompanying chemotherapy treatments.

Participants will return for each subsequent visit within a week before their next chemotherapy infusion as long as they are able to safely continue the exercise protocol. The NIRS device will be secured to the participant's leg similar to the first visit and the participants will put on the mask to measure ventilation. Participants will begin pedaling for a warmup at 0 watts for 2 minutes. After the two-minute warm up period is completed, the power output will increase to the previously calculated wattage of 1.1x LT. The participant will cycle at a self-selected cadence at this power wattage for a duration of 2 minutes ("on-kinetics"). At the end of each on-kinetics stage, participants will be asked to rate their level of effort during exercise, Rate of Perceived Exertion (RPE). The participant will then stop pedaling and will remain in recovery, sitting on the bike for 2 minutes ("off-kinetics" stage). With 5 seconds remaining in the "off-kinetics" stage, the participant will start pedaling at the same self-selected cadence for their next "on-kinetics" stage, followed by another 2-min "off-kinetics" period. This cycle of exercise followed by rest, known as on-off kinetics, will repeat for a total maximum of 3 times, or until the participant reaches volitional fatigue.

The investigators will be administering MoCA, BFI, Physical Activity Intake, PROMIS Global Health, and GLTPAQ surveys prior to participant engagement in cycling exercises. The investigators will also be administering BFI, PROMIS Global Health, and Physical Activity Follow-up surveys after each individual study session to assess changes in cancer related fatigue associated with chemotherapy treatment that may develop throughout the study time period.

Participants will undergo routine, standard of care blood draws for a CBC and metabolic testing per their managing physician with an additional tube, during the same venipuncture, for a study covered aliquot for biomarkers related to mitochondrial health for correlative research.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer or gynecological cancer without distance metastasis
* Able to perform exercise on a stationary cycle ergometer at moderate intensities for a maximum of 15 minutes
* Hemoglobin values greater than 10 at baseline
* ALT and AST values less than 2.5X the upper limit of normal by institutional standards
* Godin-Shepard Leisure time Physical Activity Questionnaire (GLTEQ) score of 14 or greater will be included. A score of less than 14 is considered insufficiency active/sedentary

Exclusion Criteria:

* Metastatic breast or gynecological cancer
* Clinically advanced cardiovascular disease
* Clinically advanced pulmonary disease
* Disease requiring continuous oxygen supplementation
* Greater than 2 centimeters or more of subcutaneous adipose tissue on the anterior thigh
* Inability to walk or stand
* Movement disorders
* Spinal cord injuries
* Autoimmune disorders
* Pregnant or breastfeeding
* Mini-Mental State Examination (MMSE) <24

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on breast cancer or gynecological cancer patients who will undergo a standard of care chemotherapy treatment as directed by their oncologist.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Muscle mitochondrial oxidative capacity | From enrollment to the end of chemotherapy treatment, an average of 12 weeks
  Study staff will measure O2Hb, HHb, and TSI, via the NIRS PortaMon device during the on-off kinetics protocol.

SECONDARY OUTCOMES:
Whole body oxygen uptake via indirect calorimetry | From enrollment to the end of chemotherapy treatment, an average of 12 weeks
  We also will measure ventilatory whole-body components including O2 and CO2 via the Parvomedics metabolic cart.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Trilk, PhD, Principal Investigator — University of South Carolina School of Medicine, Greenville; Randolph Hutchison, PhD, Principal Investigator — Furman University; Larry Gluck, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health Cancer Institute, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hutchison RE, Smith S, Caudell C, Biddle S, Gluck WL, Trilk JL. Effects of chemotherapy on skeletal muscle mitochondrial oxidative capacity using near-infrared spectroscopy (NIRS): Protocol paper for an observational mixed model repeated measures design in patients with breast and gynecological cancer. PLoS One. 2025 Jun 27;20(6):e0315351. doi: 10.1371/journal.pone.0315351. eCollection 2025. PMID 40577323

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT06672497/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT06672497/ICF_001.pdf